CLINICAL TRIAL: NCT07179146
Title: A Comparison Of Dental Arch Analysis Using 3d Digital Scanning Versus Conventional Methods In Children(A Crossover Randomized Controlled Trial)
Brief Title: A Comparison Of Dental Arch Analysis Using 3d Digital Scanning Versus Conventional Methods In Children
Acronym: Arch analysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharos University in Alexandria (Other)
Responsible Party: Principal Investigator, Nehal Salman, Lecturer of Pediatric Dentistry department, Pharos University in Alexandria
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 391/05-8-2025
Record Dates: First submitted 2025-09-01; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Dental Arch Length Analysis
Keywords: Dental arch analysis

STUDY DESIGN:
Masking Description: statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Measurement (Experimental): Using brass wire and digital caliper
  Interventions: Device: Dental arch length anlysis; Behavioral: child satisfaction; Device: Dental arch length anaylsis; Device: Dental arch length analysis; Device: Dental arch length anylsis
- Digital Measurement (Experimental): Intraoral scanning using CEREC Omnicam scanner and digital models will be obtained
  Interventions: Device: Dental arch length anlysis; Behavioral: child satisfaction; Device: Dental arch length anaylsis; Device: Dental arch length analysis; Device: Dental arch length anylsis

INTERVENTIONS:
Device: Dental arch length anlysis — Arch length
Behavioral: child satisfaction — Frankel rating scale
Device: Dental arch length anaylsis — Intermolar width
Device: Dental arch length analysis — Intercanine width
Device: Dental arch length anylsis — Arch depth

SUMMARY:
A crossover study will be conducted on 20 pediatric patients aged 7-11 years. For each participant, the upper and lower study models will be processed using two methods: the conventional method, which involves alginate impressions, and the digital method, which utilizes a 3D intraoral digital scanner (CEREC Omnicam scanner or equivalent). Measurements of arch length, arch width, and arch depth will be taken from both model types using the conventional method with a brass wire and a digital caliper. At the same time, in the scan cast, they will be calculated digitally by 3D shape software. Statistical analysis will be done to compare the results of both methods.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Children aged 7-11 years old (ASA 1).
2. Class I with normal development of occlusion .
3. Absence of dental extractions.
4. Absence of previous removable or fixed orthodontic treatments.
5. Patients with fully erupted permanent first molars.
6. Children with Frankel behavioral rating scale 2,3 and 4.

Exclusion Criteria:

1. Delayed erupted 1st permanent molar.
2. Teeth with severe rotation.
3. Dental agenesis.
4. Oligodontia.
5. Frankel behavioral rating scale 1.
6. Patients with special health care and medically compromised patients.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Subjective outcome | 2 months
  Patient acceptance will be recorded according to Modified Facial scale modified from the Maunuksela et al scale showing the 3 schematic faces representing: (A) satisfaction; (B) indifference; and (C) dissatisfaction, respectively.
Objective Outcome (Measurement) | 2 months
  arch width (inter canine and intermolar width) measured in mm
Patient acceptance | 2 months
  Frankl's behavior rating scale will be re-evaluated after each method used. Score 1-4. score 1=definitely positive, score 2=positive,score 3=negative,score 4=definitely negative.
Objective Outcome (Measurement) | 2 months
  Arch Length measured in mm
Objective Outcome (Measurement) | 2 months
  Arch depth measured in mm

CONTACTS AND LOCATIONS:
Locations (1):
- Pharos University in Alexandria, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided